CLINICAL TRIAL: NCT00405795
Title: Envision® Surface Evaluation for Patients With Stage II, Stage III, or Stage IV Pressure Ulcers
Brief Title: Envision® Surface Evaluation
Status: Completed | Type: Observational
Sponsor: Hill-Rom (Industry)
Responsible Party: Gordon MacFarlane, PhD, Director Clinical Research, Hill-Rom
Other Study IDs: MR-2005-083
Record Dates: First submitted 2006-11-28; First posted 2006-11-30 (Estimated); Last update posted 2008-07-04 (Estimated); Status verified 2008-07

CONDITIONS: Pressure Ulcer
Keywords: Pressure Ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Envision® Patient Support System

SUMMARY:
This observational study will acquire initial clinical practice utilization and product safety data for the Envision® surface.

DETAILED DESCRIPTION:
This is a single site, open label, observational study to acquire initial clinical practice utilization information, product safety, and wound healing data, as defined by changes in wound volume and/or surface area, for patients with pressure ulcers placed on this surface.

ELIGIBILITY:
Inclusion Criteria:

* Subject Weight < 400 lbs. Subject has Stage II, III, or IV pressure ulcer on weight bearing aspect of the body Subject estimated length of stay at least 7 days Subject Ability to provide informed consent

Exclusion Criteria:

* Inability to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-06; Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Levy, MD, Principal Investigator — Levindale hebrew Geriatric Center and Hospital; Cathie Papantonio, RN,BSN,CWCN, Study Director — Levindale Hebrew Geriatric Center and Hospital
Locations (1):
- Levindale Hebrew Geriatric Center and Hospital, Baltimore, Maryland, United States